CLINICAL TRIAL: NCT04754906
Title: Analysis of Motor Skills in Subjects Aged 55 and Over: the Role of Cognitive Abilities for Planning Movement.
Acronym: Vieillissement
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MANCKOUNDIA 2018
Record Dates: First submitted 2020-10-06; First posted 2021-02-15 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Mild Cognitive Disorder
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- young neurotypical subjects: people from 18 to 40 years old
  Interventions: Other: Sequence 1; Other: Sequence 2; Other: Sequence 3
- elderly neurotypical subjects: people over 55 years of age
  Interventions: Other: Sequence 1; Other: Sequence 2; Other: Sequence 3
- Elderly subjects with mild cognitive impairment: people over 55 years of age, with a diagnosis of mild cognitive impairment
  Interventions: Other: Sequence 1; Other: Sequence 2; Other: Sequence 3

INTERVENTIONS:
Other: Sequence 1 — perform arm movements towards a target
Other: Sequence 2 — judge the verticality of an object
Other: Sequence 3 — In standing position, point as quickly as possible with the right arm at the diode that will light up in front of the participant.

SUMMARY:
Falling is an event that is more frequent and severe in older age. It can lead to a loss of autonomy and a decrease in quality of life. It is therefore important to understand this phenomenon in order to better prevent it. Among the multiple risk factors associated with falling, recent research has shown a link between the decline in cognitive abilities (i.e., the mental processes that form our knowledge, such as memory) and the risk of falling. However, the impact of this cognitive decline on motor skills is still poorly understood. The purpose of this research is to study how the changes induced by aging affect motor skills. This would make it possible to take a new look at the phenomenon of falls occurring in the elderly and, in the long term, to improve the prevention and rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Neurotypical subjects group:

   * Person aged 18 to 40 years
   * Person who has given oral consent
   * Affiliated to national health insurance
   * Right-handed person
2. Group of elderly neurotypical subjects:

   * Person over 55 years of age
   * Person who has given oral consent
   * Affiliated to national health insurance
   * No cognitive problems (MMSE score >26)
   * Right-handed person
3. Elderly mild cognitive disorder subject group:

   * Person over 55 years of age
   * Person who has given oral consent
   * Diagnosis of Mild Cognitive Disorder made by a neurologist at the Centre Mémoire Ressources et Recherche (CMRR) of the University Hospital of Dijon, following the recommendations of the National Institute for Aging and Alzheimer's Association (Albert et al., 2011) This diagnosis is based on psychometric tests, brain imaging and the evolution of cognitive disorders, including an MMSE test.
   * Right-handed person

Exclusion Criteria:

* Neurological or psychiatric history with the exception of the TCL group.
* Follow-up of drug treatment in the last three months that may affect cognitive and/or motor skills.
* Received a shoulder prosthesis on the dominant side.
* Received a hip and/or knee replacement less than a year ago.
* Disabling joint disease of the hip or knee shoulder
* Protected adults (curatorship, guardianship)
* Person deprived of their liberty b judicial or administrative decision
* Pregnant, parturient or breastfeeding woman
* Major unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: young subjects, elderly neurotypical subjects and elderly subjects with mild cognitive disorder
Sampling Method: Non-Probability Sample
Enrollment: 684 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Sequence 1: symmetry ratio of the finger speed profile | through study completion, an average of 3 years
Sequence 2 : perception bias (error in degrees of angle) of dynamic subjective visual vericality | through study completion, an average of 3 years
Sequence 3 : activation time of the focal muscles in relation to the postural muscles | through study completion, an average of 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No